CLINICAL TRIAL: NCT06762795
Title: The HIEnome Study: Genome Sequencing for Perinatal HIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Seema Lalani, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-54168
Record Dates: First submitted 2024-12-20; First posted 2025-01-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn; Hypoxic Ischemic Encephalopathy; Hypoxic Ischemic Encephalopathy (HIE)
Keywords: Hypoxic-ischemic encephalopathy; Genetic testing; Genome sequencing
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perinatal HIE (Experimental): Newborns diagnosed with moderate or severe perinatal hypoxic-ischemic encephalopathy (HIE) who are undergoing therapeutic hypothermia will receive genome sequencing to identify co-morbid genetic conditions. Participants' genetic data will be analyzed for copy number variations (CNVs), single nucleotide variants (SNVs), and triplet repeat disorders per ACMG reporting standards.
  Interventions: Genetic: Genome sequencing

INTERVENTIONS:
Genetic: Genome sequencing — Neonates enrolled in this study will undergo genome sequencing with parental controls as applicable.

SUMMARY:
Perinatal hypoxic-ischemic encephalopathy is a rare severe condition in which neonates present with encephalopathy and a clinical history suggestive of prenatal or perinatal hypoxic-ischemic injury. Emerging evidence suggests that genetic conditions are frequently identified in cases of perinatal HIE; however, it is unclear which neonates with this diagnosis warrant genetic testing. This study will offer clinical genome sequencing to neonates with HIE who are undergoing total body cooling (therapeutic hypothermia) and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Delivery ≥35w0d gestation
* Diagnosed with moderate or severe HIE, or HIE with seizures
* Undergoing total body cooling / therapeutic hypothermia
* Able to provide blood or buccal samples during birth hospitalization
* Admitted to Texas Children's Hospital Main, West, or Woodlands NICU

Exclusion Criteria:

* Parents/family not willing to allow participation
* Inability to collect sufficient neonatal blood samples (in some circumstances, a buccal swab may be used as backup)

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 18 months
  The primary outcome will be the number of cases with a pathogenic or likely-pathogenic variant associated with encephalopathy. This will further be stratified by the presence or absence of a perinatal hypoxic insult or sentinel event.

SECONDARY OUTCOMES:
Genome versus exome sequencing | 18 months
  A secondary outcome will be the incremental improvement in genome sequencing versus simulated exome testing. Diagnostic variants will be classified by their genomic location: exonic, intronic, or deep intronic. The rate of diagnostic findings in genomic locations that would be assayed by exome sequencing will be compared to the overall diagnostic rate (including variants in intronic regions that would not be detected on exome sequencing) to determine the incremental diagnostic benefit of genome sequencing over exome sequencing in this population.
Indeterminate results | 18 months
  A secondary outcome will be the identification rate of non-diagnostic / indeterminate results in genes linked to conditions with an overlapping neuromuscular or neurodevelopmental phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No